CLINICAL TRIAL: NCT00033046
Title: Safety Evaluation of Cocaine Treatment Medication Modafinil: Interactions With Intravenous Cocaine
Brief Title: Evaluation of Modafinil as a Cocaine Treatment Medication and Interactions With Cocaine - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0002-1; NCT00024752 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2004-05

CONDITIONS: Cocaine-Related Disorders; Drug Administration Schedule; Infusions, Intravenous
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of this study is to evaluate modafinil, a cocaine treatment medication, and its interactions with intravenous (IV) cocaine.

DETAILED DESCRIPTION:
Placebo-controlled, escalating dose drug interaction study using a total of 12 cocaine users at a single site. Study duration will include four infusion sessions: 1) screening/baseline; 2) baseline; 3) 400mg/day steady-state modafinil; 4) 800 mg/day steady state modafinil. Infusion session will be 2 days in duration.

ELIGIBILITY:
Inclusion Criteria:

Dependent on cocaine; non-treatment seeking; male or female; DSM-4 criteria for cocaine abuse or dependence; at least 18 years of age but no older than 45 non-pregnant females using adequate birth control; capable of providing written informed consent; able to comply with protocol requirements.

Exclusion Criteria:

Additional criteria available during screening at the site

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2001-06; Study Completion 2002-04

PRIMARY OUTCOMES:
pharmacokinetic parmaters at steady state
BP, HR

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malcolm, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States